CLINICAL TRIAL: NCT06573970
Title: Atomoxetine Effect on Attention, Executive Function, and Quality of Life in Veterans With Posttraumatic Stress Disorder
Brief Title: Atomoxetine and Executive Function in PTSD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4823-R; I01 RX004823-01A2 (Other Grant/Funding Number: VA RRD)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Posttraumatic Stress Disorder With Attention Defic
Keywords: PTSD; ADHD; Executive function; Quality of life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: The study is a standard placebo-controlled, double-blind clinical trial. Within each stratum, participants will be block randomized with random block sizes of 2 and 4. Participant age and sex are randomization stratum and should retain balance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- active atomoxetine (Experimental): Active ATX (40mg capsules) will be prepared. Initial dose is 40mg, titrated to 80mg if tolerable in one week.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): placebo pill appears like real atomoxetine pill but has no therapeutic ingredient and benefit. The same schedule to distribution as Atomoxetine arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine is a selective norepinephrine reuptake inhibitor medication used to treat attention deficit hyperactivity disorder (ADHD), and executive dysfunction. Dispensing of blinded medication (40mg to 80mg ATX or placebo) will begin at randomization and will be dispensed at weeks 2, 4, 8, and 12. The initial dose of ATX is 40mg or placebo and will be given for one week, the dose will be titrated to 80mg if tolerated in the second week through week 12.
  Other Names: Strattera
  Arms: active atomoxetine
Drug: Placebo — placebo pill appears like real atomoxetine pill but has no therapeutic ingredient and benefit. The same schedule to distribution as Atomoxetine arm.
  Arms: Placebo

SUMMARY:
Attention deficits (AD) frequently co-occur with posttraumatic stress disorder (PTSD). The presence of AD is associated with greater PTSD clinical severity and poorer clinical outcomes. Knowledge regarding the mechanism underlying this association is limited, though the emerging evidence has indicated that executive function deficit (EFD) is strongly correlated with AD and PTSD symptoms. While treatments developed for PTSD have existed for years, a substantial portion of individuals do not fully respond to conventional treatment. Accumulating evidence suggest that attention deficit (AD) and EFD may be a driving force for PTSD treatment resistance. However, treatment of executive impairment in PTSD is very limited. As a result, untreated co-occurring AD and EFD in PTSD poses severe negative impacts on patients' functional recovery, treatment outcomes, and quality of life (QoL). Given that up to 50% of patients do not respond well to the first-line pharmacological PTSD treatments, it is imperative to seek novel treatment strategies to improve EF that may improve both standard treatment response and QoL, social function. The proposed study directly addresses this knowledge gap by testing the efficacy of atomoxetine (ATX) in improving EF and attention among Veterans with PTSD, which will further improve Veterans' QoL and social function. ATX represents a promising novel candidate pharmacotherapy for individuals with PTSD. ATX is a non-stimulant selective norepinephrine reuptake inhibitor (SNRI), approved by the FDA for the treatment of ADHD. Studies suggest that ATX, unlike stimulants, lacks addictive properties and shows efficacy in the treatment of comorbid depression and anxiety, which is ideal in the treatment of PTSD. Data from the investigators' preliminary study provides encouraging support for the therapeutic potential of ATX in improving EF in Veterans with comorbid PTSD/ADHD. The investigators' recent research uncovered a higher rate of ADHD among Veterans with PTSD, and the comorbid AD symptoms were correlated with PTSD severity and poorer treatment outcomes. Treatment with ATX showed significant symptoms reduction in ADHD and improvement in inhibitory function in Veterans with ADHD/PTSD. In the proposed study, the investigators will focus on ATX in improvement of EF and attention, and further psycho-social life function and QoL. The investigators will (1) employ a randomized, double-blind design that will consist of 12 weeks of treatment with ATX or placebo medication; (2) use standardized, repeated dependent measures to rigorously assess AD and EFD symptomatology; (3) measure impairment in associated mental and behavioral health problems (e.g., attention deficit, depression, anxiety, suicidality, QoL, family/social functioning); and (4) use response inhibition task GoNogo, working memory and attention tests Digit Span and Trail Making to investigate the underlying pathophysiology of PTSD and prognostic indicators of treatment outcome. To achieve these goals, the investigators have assembled a multidisciplinary team with expertise in PTSD, ADHD clinical trials, and human laboratory paradigms who have successfully collaborated in the past and are uniquely qualified to implement this type of investigation. The proposed project is directly responsive to the mission of the VA-RRD "to maximize Veterans' functional independence, quality of life and participation in their lives and community." Successful completion of this study will provide a platform for a large multi-center trial to further confirm the important role of EF in PTSD treatment outcomes. The findings from this study will provide critically needed evidence to help inform clinical practice guidelines on the treatment of PTSD. The outcome of the proposed research will be significant, because it provides a knowledge base to allow for development of new PTSD intervention strategies. More importantly, this clinical trial may immediately benefit Veterans by enhancing their cognitive function, reducing AD related disability, and further improving quality of life for Veterans who suffer from PTSD.

DETAILED DESCRIPTION:
Aim 1: To examine the impact of ATX in enhancing executive function. Based on preliminary data, the investigators hypothesize that ATX, compared with placebo, will be more effective in improving EF in Veterans with PTSD and AD. To test this hypothesis, 12-week, randomized, double-blind, placebo-controlled trial of ATX will be conducted among Veterans with PTSD. The outcome measure will be the analyses of changes in Behavior Rating Inventory of Executive Function-Adult (BRIEF-A), the response inhibition task, GoNogo (GNG), Trail making and digit span tests (TMT and DST). The rationale for this aim is that impaired EF may be a powerful risk for PTSD treatment resistance and poor QoL and psychosocial function (PSF), therefore, improving EF with ATX may ultimately improve Veterans QoL, PSF, and reducing disability rating. The investigators expect that the 12-week treatment with ATX will significantly improve attention, EF, inhibitory function in Veterans with PTSD.

Aim 2: To examine the impact of ATX on improvement of QoL and daily psycho-social function.

Based on literature and preliminary data, the investigators hypothesize that ATX, compared with placebo, will be more effective in improve Veterans' QoL, PSF, and disability rating. The outcome measure will be the analyses of changes in Adult ADHD Quality of Life-29 (AAQOL-29), WHO Disability Assessment Schedule 2.0 (WHODAS 2.0), The Inventory of Psychosocial Functioning (IPF). The investigators expect that the 12-week treatment with ATX will significantly improve QoL and psychosocial function, and significantly reduce EFD and AD related disability.

Aim 3: To examine the impact of ATX on overall AD and PTSD treatment outcomes. The hypothesis for this aim is that successful treatment of attention and executive deficits will be associated with greater reduction of PTSD and AD symptoms. To achieve this goal, more clinical and psychological assessments including depression, anxiety, and other functional scales, such as CAPS-5 scores, BDI, BAI, and CARRS-S:S attention deficit scores will be performed to assess the PTSD overall improvement. The investigators expect that the significant improvement of attention and executive function will lead to a significant improvement of overall PTSD outcomes.

Recruitment:

Recruitment of subjects will take place in three sites, including the Ralph H. Johnson (RHJ) VAMC, Savannah VA Community Based Outpatient Clinic (CBOC), and Hinesville CBOC. The decision to use three sites were based on the calculation of study sample size, the availability of the target patient population, and the feasibility of recruiting the proposed study sample.

The investigators will devote 2 months to study start-up; 40 months for active recruitment (10 months in year 01, 12 months in year 02 and year 03, 6 months in year 04); 3 months for the patients enrolled in the last recruitment month to complete the treatment and follow-up; 1 months for the study close-out; and 6 months for data analysis. The total length of study will be 4 years. The investigators plan to recruit 160 subjects with PTSD in 4 years, and allow 20% dropout with a final of 128 subjects (64 from the RHJ VAMC, 32 from the Savannah CBOC, and 32 from the Hinesville CBOC) entering to the final analysis.

The investigators plan to recruit subjects seeking outpatient treatment in the VA PTSD Clinician Team (PCT) clinics and the Mental Health Service Line (MHSL) clinics at RHJ VAMC, and at Savannah and Hinesville CBOCs. The primary source of recruitment will be PCT clinic referrals by PCT intake team, which also referring patients to Savannah and Hinesville clinic. As the PI and coinvestigators in this research project are either directors or attending physicians in each of the three sites, the investigators will have direct contact with patients assigned to the PCT clinics and MHSL clinics. Therefore, the investigators anticipate no difficulty in recruiting 1 PTSD subject every 2 weeks from RHJ VAMC, and 1 PTSD subject/4weeks from each of the CBOCs. This estimate is very reasonable, as the investigators recruited over 44 subjects in 2 years in the Preliminary Study only at RHJ VAMC. In the investigators' previous studies, it was found about 50% of Veterans with PTSD meet the ADHD criteria (Adams et al, 2015). Flyers will also be posted in appropriate areas of VAMC facilities.

Treatment Duration:

The double-blind treatment will last 12 weeks. Study visits will be scheduled at weeks 2, 5, 9, and 13. Safety assessment, such as C-SSRS will be conducted at each visit. In addition, the C-SSRS will also be conducted by weekly phone call between in-person visits. Patients randomized after the initial assessment. Those patients will be followed until the end of the study. Following their final visit, subjects will be referred to their primary care physician for a clinical follow up treatment. The 4th treatment visit and final follow up visit can both be virtual if the subjects chooses to do so, this decision will be optional depending on the subject's preference.

Data Collection:

An operations manual and case report form will be developed. The site study coordinator will collect all data. After a patient consent to participate in the study, the site coordinator will create a patient casebook, which will contain the consent forms, all relevant source documents, and any other information pertinent to the study. The case report forms will be completed at each visit. This is a password-protected system that is accessed through the VA intranet. The study personnel, including the biostatistician, statistical programmer, database programmer, will have access to read the data. The information collected about the patients during the course of the trial will be stored at the Research Database Storage in the Charleston VAMC PTSD Program. The database will be shared among the researchers involved in this project in the future, but information that would disclose personal identity (name, address, telephone, and security number) will not be released and will always be kept separate from the research database.

Primary Data Analysis:

Baseline clinical and demographic characteristics will be collected, and association of baseline characteristics and clinical predictors of study outcomes will be performed utilizing appropriate regression models. Study outcomes will be collected longitudinally at study baseline, during study treatment (weeks 8, 12) and at study follow-up (week 16). Continuous study outcomes (BRIEF-A, TMT, and DST (Aim1); AAQoL, IPF, and WHODAS (Aim2); CAPS-5, and CARRS (Aim3)) will be assessed utilizing linear mixed effects regression models (LMM) including all post randomization time points. Transformations using restricted cubic splines or fractional polynomials will be considered for continuous model covariates if significant departure from linearity is detected. Normality of residuals will be assessed through Q-Q plots and when departure from normality is detected, appropriate transformations of non-parametric modeling will be utilized. Generalized linear mixed effects regression models (GLMM) will be utilized for assessment of count data (GoNoGo omission/commission errors, suggesting inattention and impulsivity). For count GoNoGo omission and commission error measures, overdispersion will be evaluated and alternative models (e.g., negative-binomial, zero-inflated) used as needed. Further, the GoNoGo task will record latency to response in the Go tasks. With the possibility of temporal trends in the longitudinal collection of data (learning) as well as non-response during the response window (fixed censoring), random effects survival models will be considered to examine study group differences in response time (RT) to Go tasks. Contrasts of interest (end of treatment outcomes) will be assessed with model based least square means and associated standard errors. Subgroup analyses will be pre-specified and considered exploratory. Treatment heterogeneity by clinic will be evaluated using appropriate models with clinic-by-treatment interaction. Both naïve and adjusted models will be presented; naïve models will contain design specific covariates only (study visit, baseline response, study clinic, and treatment assignment when appropriate) while covariate adjusted models will be developed using characteristics that were found to be significantly associated with study outcomes or are previously known confounders. In all longitudinal models, a treatment by time interaction will be included to assess differential response over the course of study treatment and when found significant, stratified analysis will be performed and results presented. Participants positively responding to all Go and NoGo tasks will be assessed for task compliance on a per participant basis. Sensitivity analysis with and without participant data will be conducted to assess the impact of such instances, although the investigators expect the occurrence rate to be minimal. To assess the synchronous relationship between primary study outcomes and cooccurring measures of depression and anxiety, time varying covariates (BAI, BDI) will be independently added to each model and assessed for significance. Further, moderation of outcomes by both baseline, and concurrent measures of depression and anxiety will be evaluated through model interaction terms (ATX x depressions/anxiety). When significant, stratified analysis will examine the relationship between depression and anxiety with each outcome and compared across treatment groups.

Secondary Data Analysis:

To assess if improvements in EF during study treatment are associated with co-occurring QoL, IPF, PTSD and AD symptom improvement, LMM will be developed including the time varying effect of EF variables (BRIEF-A, GNG) on QoL, WHODAS, IPF) and on PTSD (CAPS-5) as well as AD symptoms (CARRS). At each treatment measurement timepoint, change from study baseline will be calculated as a summary measure prior to analysis. Both concurrent and time lagged independent variables will be assessed for association. Following completion of the primary analysis described above, durability of treatment efficacy will be performed on measured collected at the study follow-up visit. Similar linear and generalized linear models will be developed to assess outcomes as described in the primary data analysis section.

Missing Data:

Missing data in longitudinal studies can be a problematic feature but can be mitigated through study design considerations. To minimize missing data and study attrition, study simplification and enhanced communication between study coordinators and participants will be emphasized. The investigators will make every effort to prevent attrition, e.g., telephone reminders prior to visits, participation compensation, flexible scheduling, and reinforcing adherence at each visit. However, these methods do not ensure that all data will be collected, and appropriate analytic methods will be employed to accommodate missing data (e.g. multiple imputation). In addition, in keeping with the ITT principal, the investigators will make every effort to continue assessments for the entire course of randomized treatment, even among those who stop participating in the study assigned intervention or fail to complete the full medication time course.

Data Quality Assurance:

REDCap facilitates the process of gathering and storing data, ensuring proper documentation of variables, checking data validity, and facilitating the processes of creating analytic databases for statistical analyses. For each variable, a set of range and consistency checks will be developed by the biostatistician in conjunction with the Principal Investigator and Research Coordinator. Data will be audited for correctness by two independent data-entry personnel periodically (quarterly) and discrepancies will be evaluated, and any errors identified will undergo review and resolution. Data ranges will be assessed, and examination of outliers performed during quarterly data checks. Extreme values that are plausible will be retained in the analysis. Implausible data will be flagged for additional checks (ie. a report of 500 cigarettes smoked per day).

Data and Safety Monitoring:

The data safety monitoring committee (DMC) will be charged with monitoring this proposed clinical trial. This DMC will be constituted specifically for this study. The DMC will provide ongoing independent evaluation of the study progress including participant accrual and retention, adverse events monitoring, and data analysis plan. The DMC will be comprised of a minimum of three experts in clinical research including an internal medicine physician, a psychiatrist, and another clinical scientist with statistical expertise. The DMC will initially meet before study start-up and at that time will determine the frequency of subsequent reviews. It is proposed that the DMC meet at least every 6 months. In addition to the above noted safety and accrual parameters, the DMC will also review completeness of follow-up, data quality, protocol deviations, and review protocol modifications. Within each DMC report, balance of important study characteristics will be assessed across blinded study groups (A/B); specifically race/ethnicity, baseline PTSD and AD measures. Participant age and sex are randomization stratum and should retain balance, however, these will also be assessed at each DMC meeting.

Dosing Schedule: The medication (40mg to 80mg ATX or placebo) schedule is shown in Table 3. Dispensing of blinded medication will begin at randomization and will be dispensed at weeks 2, 4, 8, and 12. The initial dose of ATX is 40mg or placebo and will be given for one week, the dose will be titrated to 80mg or placebo daily if tolerated in the second week through week 12.

Medication Packaging, Assignment and Dispensing Plan:

Active and placebo ATX (40mg capsules) will be designed by Dr. David Shirley at the Plantation Pharmacy, Charleston SC, then labeled, packaged, and distributed by the VA Clinical Research Pharmacy Coordinators. Packaging will consist of boxes containing either ATX or placebo. For the active treatment periods, capsules will be boxed to contain a four-week supply. Each box will be uniquely numbered, and the box numbers will be tied to their contents (active or placebo) in a database at the Charleston VAMC. This database will also contain the randomization treatment assignment of each participant. At each dispensing visit site, personnel will access via a password - secured Kit Assignment Program on the study's SharePoint website to obtain box numbers for dispensing to a specific participant. To ensure that each patient is assigned boxes filled with capsule corresponding to their treatment assignment, all blinded box assignments will require the use of two unique patient identifiers. Records will be maintained of all doses dispensed, and Veterans will be asked to return all unused tablets and empty prescription vials to the clinic for assessment of treatment compliance.

Assessment of Compliance and Methods to Maximize Compliance:

Medication will be stored and dispensed from the VAMC investigational drug pharmacy. Records will be maintained of all doses dispensed, and Veterans will be asked to return all unused tablets and empty prescription vials to the clinic for assessment of treatment compliance.

Compliance with medication will be assessed via returned capsule count in the presence of the patient at each visit, which is a traditional method of compliance assessment. Methods successfully utilized to help minimize study withdrawals, including follow-up phone calls, and availability of 24-pager coverage to discuss medication-related and other issues, will also help maximize medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* Veterans ages 18 to 75 with PTSD and AD (CAPS > 35 for age 18 to 64, CAPS > 25 for age 65 to 75; CAARS-S:S > 60)

  * The cut-score of 25 used for participants age 65 to 75 because lower cut-score has been recommended for older Veterans (Yeager and Magruder, 2014)
  * ADHD has been recognized as a neurobehavioral impairment in executive function (Brown, 2008)
  * Veterans with PTSD at this age range are suited for this study because statistically they have fewer confounding variables for this clinical trial, including medical conditions such as hypertension or glaucoma and cognitive impairments such as dementia
* Physical health good enough to be able to participate in the study
* Competent to give informed consent

Exclusion Criteria:

* Age younger than 18 or greater than 75

  * Age becomes the main risk factor for major neurocognitive disorder, especially after 75 (Sousa et al, 2020)
* Known sensitivity to ATX
* Presence of disorders that could conceivably be exacerbated by atomoxetine

  * specifically, narrow angle closure glaucoma, urinary outflow obstruction, hypertension, and neurological disorders, particularly tics and Tourette's syndrome, or a history of epilepsy or seizures
* Subjects with major traumatic brain injury (TBI) determined by Ohio State University Traumatic Brain Injury Identification Method (OSU-TBI ID)
* However, mild TBI, assessed with OSU-TBI ID and review of record will be allowed to participate in this trial
* Use of concomitant medication that could potentially interact with atomoxetine including monoamine oxidase inhibitors (MAOI), antihypertensive medication, or any concomitant medication that is a cytochrome 2D6 (CYP2D6) inhibitor, such as paroxetine, venlafaxine, fluoxetine, because atomoxetine's elimination involves the CYP2D6 system
* Subjects who are currently taking psycho-stimulants, other NRIs such as duloxetine, and venlafaxine will be excluded

  * However, the investigators will allow subjects who stopped the psycho-stimulant or other NRI or other SSRIs 2 weeks prior to the start of the trial
* Subjects receiving active ongoing therapy with good response at the point of recruitment

  * The project will allow approved standard therapies, including psycho- or/and pharmacotherapies be continued with the condition that the subjects continue to present with PTSD symptoms severe enough to meet the inclusion criteria
* An active or lifetime major mental health diagnosis as determined by DSM-5 major psychiatric disorders, including:

  * schizophrenia
  * schizoaffective disorder
  * psychotic disorder not otherwise specified
  * bipolar I disorder, bipolar II disorder
  * bipolar disorder not otherwise specified

    * The project will allow the presence of depressive disorders if the depressive episodes are secondary to PTSD
* Current substance use disorders:

  * DSM-5 alcohol
  * marijuana
  * and/or other drug use disorders in the last 3 months

    * Mild alcohol and marijuana use which does not meet the criteria for mild use disorder, such as occasional or recreational use will be permitted on a case by case basis
* Females who are pregnant or desired to become pregnant during the clinical trial period

  * Urine pregnancy tests will be performed at each of the visits, including prior to, during, and after the clinical trial
* Prominent suicidal or homicidal ideation or any suicidal behavior in the past 3 months on the Columbia Suicide Severity Rating Scale (C-SSRS)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-06-29 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function-Adult (BRIEF-A) | 15 minutes
  The BRIEF-A is a 75-item questionnaire that assesses adult executive functioning and self-regulation. It's suitable for adults ages 18-90 with a wide range of developmental, neurological, psychiatric, and systemic disorders. BRIEF-A uses a 3-point scale to rate items on a frequency basis, with 0 indicating "never", 1 indicating "sometimes", and 2 indicating "often". The raw scores, range from 0 to 150, of each scale are added together to calculate T scores. The higher T scores reflecting greater degree of executive dysfunction and levels of impairment, with scores at or above 65 suggestive of clinical significance.

SECONDARY OUTCOMES:
Conners' Adult ADHD Rating Scales-Self Report: Short Version (CAARS-S:S) | 10 to 15 minutes
  The CAARS-S:S is a 26-item self-report screening measure assessing the extent to which one experiences ADHD symptoms and related problems. The CAARS S:S generates an ADHD Index and four factor-derived subscales; (1) Inattention/Memory Problems, (2) Hyperactivity/Restlessness, (3) Impulsivity/Emotional Lability, and (4) Problems with Self-Concept. Raw scores were converted to t-scores using age- and sex-normative data. The raw scores range from 0 to 78, Higher scores on the subscales indicate greater presence of self-reported ADHD-related characteristics. T-scores above 65 indicate a likelihood of moderate to severe ADHD symptoms and impairment.
Clinician Administered PTSD Scale 5 (CAPS-5) | 20 minutes
  The CAPS-5 is a 30-item structured interview that assesses both target PTSD symptoms and impact of symptoms on social and occupational functioning. The CAPS-5 is the gold standard for diagnosing PTSD. It provides both a dichotomous index for PTSD diagnoses and PTSD symptom severity. CAPS-5 has a total score range of 0-80. This score is calculated by adding the individual severity scores (0-4) for each of the 20 PTSD symptoms. Higher scores indicate more severe PTSD symptoms.

OTHER OUTCOMES:
The Adult ADHD Quality of Life-29 (AAQOL-29) | 15 minutes
  AAQoL-29 is a 29-item scale measures health-related quality of life (QoL) in adults with ADHD. The AAQoL produces a total score and four subscale scores: Life Productivity, Psychological Health, Life Outlook, and Relationships. The AAQoL items are rated on a five-point Likert scale, with 1 indicating "Not at all/Never" and 5 indicating "Extremely/Very Often" with a total score from 29 to 145. A higher score indicates a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhewu Wang, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
As this is a single site study and all data analysis will be completed at the primary site (Charleston). All collected clinical, demographic, and geographic data, as well as treatment data will be stored in Charleston VAMC clinical trial data bank. This study is led by PI, Dr. Wang, and Co-Investigators, Drs. Hamner, Acierno. Both PI and co-Investigators will have access to the data. They will be involved in the data analysis and in interpretation of the data results. Also, the biostatistician, Mr. Baker will further contribute to the data analysis and validation.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Records will be maintained and destroyed per the VHA Records Control Schedule (RCS 10-1). The paper data collected from this study will be kept in a locked cabinet in a locked office, while the electronic data will be coded and stored without personal identifiers. The data will be available from January 2025 until 6 month after the trial completion.
Access Criteria: The Investigator will make study data accessible to the monitor, other authorized representatives of the Sponsor (or designee), IRB/IEC, and Regulatory Agency (e.g., FDA) inspectors upon request. A file for each subject must be maintained that includes the signed Informed Consent, HIPAA Authorization and copies of all source documentation related to that subject.